CLINICAL TRIAL: NCT00596102
Title: Longterm Immunogenicity of the Japanese Encephalitis Vaccine IC51. An Uncontrolled Phase 3 Follow-up Study
Brief Title: Longterm Immunogenicity of the Japanese Encephalitis Vaccine IC51
Status: Completed | Type: Observational
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: IC51-303
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-06

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Observational Model: Cohort

INTERVENTIONS:
Biological: Japanese Encephalitis purified inactivated vaccine — Japanese Encephalitis purified inactivated vaccine

SUMMARY:
The study investigates the long term safety and immunogenicity of the Japanese Encephalitis vaccine IC51 up to month 60.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects at least 18 years of age
* Written informed consent obtained prior to study entry
* Subjects correctly included and having completed clinical studies IC51-301 (NCT00604708) and IC51-302 (NCT00605085) with at least one vaccination

Exclusion Criteria:

* Inability or unwillingness to provide informed consent and to abide the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 3,300 subjects having completed IC51, JE-VAX or placebo treatment in studies IC51-301 or IC51-302 will take part in the safety follow up, up to month 6 after 1st vaccination in the study IC51-301 (NCT00604708) or IC51-302 (NCT00605085).
  Only ~160 subjects, who have been treated with IC51 will take part in the immunogenicity and long-term analysis up to month 60.
Sampling Method: Non-Probability Sample
Enrollment: 3258 (Actual)
Dates: Start 2005-10; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Hatzenbichler, Ph.D., Study Director — Valneva Austria GmbH

REFERENCES:
- [Derived] Taucher C, Kollaritsch H, Dubischar KL. Persistence of the immune response after vaccination with the Japanese encephalitis vaccine, IXIARO(R) in healthy adults: A five year follow-up study. Vaccine. 2019 May 1;37(19):2529-2531. doi: 10.1016/j.vaccine.2019.03.030. Epub 2019 Apr 5. PMID 30962094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study participants were recruited from 44 study centers previously participating in study IC51-301 and IC51-302
Groups:
- IC51: no active treatment in study IC51-303, IC51 vaccinations were performed in preceeding study IC51-301 or IC51-302
- JE-VAX: no active treatment in study IC51-303, vaccinations were performed in preceeding study IC51-301
- Placebo: no treatment in study IC51-303, vaccinations were performed in preceeding study IC51-302
Period: Up to Month 6
Arm/Group | IC51 | JE-VAX | Placebo
Started | 2283 | 338 | 637
Completed | 2283 | 338 | 637
Not Completed | 0 | 0 | 0
Period: Up to Month 60
Arm/Group | IC51 | JE-VAX | Placebo
Started | 2283 | 338 | 637
Completed | 102 (long-term safety follow-up beyond Month 6 for a sub-set of subjects in "IC51" group only) | 0 | 0
Not Completed | 2181 | 338 | 637

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 | JE-VAX | Placebo | Total
Number analyzed (Participants) | 2283 | 338 | 637 | 3258
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (13.8) | 42.3 (14.1) | 33.5 (13.0) | 35.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1274 | 201 | 365 | 1840
  Male | 1009 | 137 | 272 | 1418
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 38 | 1 | 16 | 55
  Black or African American | 101 | 35 | 25 | 161
  Caucasian | 2076 | 288 | 574 | 2938
  Other | 68 | 14 | 22 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Seroconversion Rate (SCR) ≥ 1:10 Anti-JEV Neutralizing Antibody Titer (PRNT)
Description: first vaccination refers to 1st vaccine administration in studies IC51-301 or IC51-302
Time Frame: 24 months after the first vaccination
Population: subjects enrolled into this study who planned to participate in the long-term immunogenicity part and received IC51 in the respective preceeding study
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | IC51
Number analyzed (Participants) | 181
percentage of subjects | 81.8 [75.7 to 86.7]

2. Secondary Outcome: Percentage of Subjects With Seroconversion Rate (SCR) ≥ 1:10 Anti-JEV Neutralizing Antibody Titer (PRNT)
Time Frame: 6, 12, 36, 48 and 60 months after 1st vaccination
Reporting Status: Not Posted

3. Secondary Outcome: Geometric Mean Titers
Time Frame: 6, 12, 36, 48 and 60 months
Reporting Status: Not Posted

4. Secondary Outcome: Adverse Events
Time Frame: 6, 12, 24, 36, 48 and 60 months after 1st vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: all participants across all treatment groups were followed-up until Month 6; a sub-group of the IC51 treatment arm was followed-up until Month 60
Description: group "IC51 Month 6" includes the sub-set of study participants that later on is followed-up until Month 60 (group "IC51 Month 60")
Groups:
- IC51 Month 6: no active treatment in study IC51-303, IC51 vaccinations were performed in preceeding study IC51-301 or IC51-302; follow-up till Month 6
- JE-VAX: no active treatment in study IC51-303, JE-VAX vaccinations were performed in preceeding study IC51-301 or IC51-302; follow-up till Month 6
- Placebo: no active treatment in study IC51-303, Plarcebo vaccinations were performed in preceeding study IC51-301 or IC51-302; follow-up till Month 6
- IC51 Month 60: no active treatment in study IC51-303, IC51 vaccinations were performed in preceeding study IC51-301 or IC51-302; follow-up till Month 60
Arm/Group | IC51 Month 6 | JE-VAX | Placebo | IC51 Month 60
Serious Adverse Events (participants affected / at risk) | 15/2283 | 2/338 | 7/637 | 14/102
Other Adverse Events (participants affected / at risk) | 78/2283 | 16/338 | 31/637 | 54/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Month 6 (N=2283) | JE-VAX (N=338) | Placebo (N=637) | IC51 Month 60 (N=102)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Appendix Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Appendiceal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia Fructure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenocarinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Central Nervous System Inflammation (Nervous system disorders) | 1 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Mediastinal Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Meniscus Operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Coronary Stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Abscess Soft Tissue (Infections and infestations) | 0 | 0 | 0 | 1
Endometritis (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Smear Cervix Abnormal (Investigations) | 0 | 0 | 0 | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Toe Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Urethral Stricture (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Blood Donor (Social circumstances) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Month 6 (N=2283) | JE-VAX (N=338) | Placebo (N=637) | IC51 Month 60 (N=102)
Nasopharyngitis (Infections and infestations) | 78 | 16 | 31 | 19
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 10 | 0 | 3 | 3
Acute Tonsillitis (Infections and infestations) | 6 | 4 | 1 | 3
Bronchitis (Infections and infestations) | 13 | 2 | 4 | 6
Cystitis (Infections and infestations) | 11 | 0 | 3 | 7
Herpes Simplex (Infections and infestations) | 3 | 0 | 1 | 3
Pneumonia (Infections and infestations) | 4 | 0 | 2 | 3
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 3
Tonsillitis (Infections and infestations) | 6 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 17 | 2 | 6 | 4
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 3 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 1 | 3 | 3
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 3 | 3
Headache (Nervous system disorders) | 42 | 1 | 7 | 4
Depression (Psychiatric disorders) | 5 | 2 | 0 | 4
Dental Implantation (Surgical and medical procedures) | 1 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other